CLINICAL TRIAL: NCT05623995
Title: Effect of Evolocumab on Chronic Total Occlusions After Successful Percutaneous Coronary Intervention (EVOLO-CTO)
Brief Title: Effect of Evolocumab on Chronic Total Occlusions (EVOLO-CTO)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lin Zhao (Other)
Responsible Party: Sponsor-Investigator, Lin Zhao, Principal Investigator, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-22
Record Dates: First submitted 2022-11-07; First posted 2022-11-21 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: In-stent Restenosis; Major Adverse Cardiovascular Events
Keywords: Chronic total occlusion; Restenosis
MeSH Terms: interventions — evolocumab; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Participants will receive PCSK9 inhibitors added to guideline recommended statin therapy.
  Interventions: Drug: PCSK9 inhibitor
- Control arm (Active Comparator): Patients will continue to taking guideline recommended statin therapy.
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: PCSK9 inhibitor — Evolocumab per every two weeks, starting at day 1 and up to week 48, added to guideline recommended statin therapy..
  Other Names: Evolocumab
  Arms: Treatment arm
Drug: Statin — Guideline recommended statin therapy.
  Other Names: Hydroxymethylglutaryl-Coenzyme A Reductase inhibitor
  Arms: Control arm

SUMMARY:
The purpose of this study is to evaluate the effect of proprotein convertase subtilisin/kexin type-9 (PCSK9) inhibitors added to regular statin therapy on target lesion failure (TLF) and arteriosclerosis progression in patients with chronic total occlusions (CTOs) undergoing successful percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Chronic total occlusions (CTOs) are found in 15-25% of patients with stable angina pectoris. The presence of a CTO indicates unfavorable prognosis, with higher rate of major adverse cardiovascular events. Statins are frequently used after PCI in order to lower LDL cholesterol levels and reduce the chances of coronary artery obstruction recurring. Despite this preventive measure, high risk for restenosis and re-occlusion was observed a significant proportion of patients with CTOs undergoing PCI.

Proprotein convertase subtilisin/kexin type-9 (PCSK9) inhibitors represent a novel class of lipid-lowering drugs leading to rapid, profound, and consistent reductions in LDL-C levels. The effect of PCSK9 inhibitor in patients with CTO, after a recent PCI is not known.

In this study the investigators want to evaluate the effect of the PCSK9 inhibitor on neointimal hyperplasia and target lesion failure (TLF) in patients with CTOs receiving regular statin treatment. A serial of intravascular ultrasound imaging study will be performed to determine the arteriosclerosis progression at 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age with written informed consent
* Presence of a CTO in native coronary artery.
* Stable angina or myocardial ischemia in a territory supplied by CTO
* CTO located in segments 1-3 (RCA), 6-7 (LAD), 11-12 (LCx)
* Target artery ≥2.5mm
* Scheduled to undergo percutaneous coronary intervention (PCI)
* LDL-C ≥70 mg/dL (≥1.8 mmol/L) in patients who have been on any stable statin regimen for ≥ 4 weeks prior to enrollment; or LDL-C ≥125 mg/dL (≥3.2 mmol/L) in patients who are statin-naïve or have not been receiving stable statin regimen for ≥ 4 weeks prior to enrollment

Exclusion Criteria:

* Acute myocardial infarction within 1 month
* Known severe chronic kidney disease (estimated Glomerular Filtration Rate [eGFR] <60 mL/min/1.73m2 or serum creatinine level >2.5 mg/dL);
* History of allergy to iodine contrast agents
* Allergy to PCSK9 inhibitors or any other ingredients contained in study drug
* Pregnancy or breastfeeding
* Persistent or permanent atrial fibrillation
* Patients with history of coronary artery bypass graft
* Inability or unwilling to provide informed consent
* Malignant neoplasms or Major illness with life expectancy <1 year
* Planned coronary revascularization or major non-cardiac surgery 12 months after intervention
* Patients previously treated with PCSK9 inhibitors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in percent plaque volume and plaque burden. | 12 months
  Change in percent plaque volume and plaque burden by intravascular ultrasound (IVUS) between PCSK9 inhibitors group and control group.

SECONDARY OUTCOMES:
Rate of Target Lesion Failure (TLF) | 12 months
  TLF is defined as a composite of: all cardiac death, target vessel myocardial infarction (SCAI definition), and clinically driven target lesion revascularization (TLR).
Neointimal volume with intravascular ultrasound (IVUS) (mm3 per 1mm) | 12 months
  Comparison of neointima volume by IVUS between PCSK9 inhibitors group and control group.
Ischemia | 12 months
  Ischemic burden assessed with CMR from baseline to 3 and 12 months follow-up
Change in left ventricular systolic function assessed with CMR | 12 months
  The left ventricular ejection fraction assessed with CMR from baseline to 3 and 12 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Lin Zhao, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No